CLINICAL TRIAL: NCT06929039
Title: A Randomized , Open Label, Three Arm, Parallel Group, Single Dose, Comparative Pharmacokinetic , Safety, and Immunogenicity Study Comparing KSHB002 (Abatacept) 125 mg/ ml Pre-filled Injection With US-Licenced ORENCIA and EU-Approved ORENCIA Administered Through Subcutaneous Route in Healthy Adult Human Volunteers
Brief Title: Open Label , Randomized, Three Arm Parallel Group Single Dose Comparative Pharmacokinetic , Safety and Immunogenicity Study in Healthy Subjects
Acronym: abatacept
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kashiv BioSciences, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSHB002
Record Dates: First submitted 2025-01-31; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-01

CONDITIONS: Rheumatoid Arthritis (RA
Keywords: abatacept; kashiv biosciences
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Test Product (Experimental): Test Product- KSHB002 Abatacept 125mg/ml Pre-filled syringe
  Interventions: Drug: Abatacept
- Reference Product 1 (Active Comparator): US-Liceneced Orencia 125mg/ml Pre-filled syringe
  Interventions: Drug: Abatacept
- Reference product 2 (Active Comparator): EU-Approved Orencia 125mg/ml pre-filled injection
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Test Product (A) (Kashiv's Abatacept): KSHB002 (Abatacept) Injection, 125 mg/mL - Manufactured by: Kashiv Bioscience's LLC, USA.
  Arms: Test Product
Drug: Abatacept — Reference Product (B) (US-licensed ORENCIA): 'ORENCIA' (abatacept) injection 125 mg/mL - Manufactured for: Bristol-Myers Squibb Company Princeton, NJ 08543 USA.
  Arms: Reference Product 1
Drug: Abatacept — Reference Product (C) (EU-authorized ORENCIA): 'ORENCIA' 125 mg solution for injection (abatacept) - Marketing Authorization Holder: Bristol-Myers Squibb Pharma EEIG, Plaza 254, Blanchardstown Corporate Park 2, Dublin 15, D15 T867, Ireland.
  Arms: Reference product 2

SUMMARY:
The goal of this clinical trial is to learn if Test Product KSHB002 shows equivalence in terms of PK , safety and immunogenicity as compared to reference product ORENCIA used to treat Rheumatoid arthritis .

Participants will:

Take drug Test or a reference subcutaneously as a single dose and these participants will be healthy volunteers

Primary Endpoint: The following pharmacokinetic parameters will be determined as: Cmax and AUCi, of KSHB002 (Abatacept), US-licensed ORENCIA and EU-authorized ORENCIA.

Secondary Endpoint : Safety will be evaluated from occurrence of adverse events post dose. The number, severity and relation to treatment will be collected by the reporting of the adverse events (AE) and monitoring of clinically relevant changes e.g., vital signs, physical examination and lab values in blood and urine.

* Immunogenicity will be evaluated from the number/percentage of subjects positive for ADA (Anti-Drug Antibody) and Neutralizing Anti-drug antibody
* Secondary pharmacokinetic endpoints will be evaluated as AUCt, Tmax, Kel and tHalf.

DETAILED DESCRIPTION:
A randomized, open label three-arm, parallel group, single dose comparative pharmacokinetic, safety and immunogenicity study comparing KSHB002 (Abatacept) Injection, 125 mg/mL with US-licensed ORENCIA and EU-authorized ORENCIA administered through subcutaneous route in healthy adult human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or non-pregnant, non-lactating female. A. Female of childbearing potential must have a negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test at screening. They must be using an acceptable form of contraception.

B. For female of childbearing potential, acceptable forms of contraception include the following:

i. Non hormonal intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or ii. Barrier methods containing or used in conjunction with a spermicidal agent, or iii. Surgical sterilization or iv. Practicing sexual abstinence throughout the course of the study.

C. Female will not be considered of childbearing potential if one of the following is reported and documented on the medical history:

i. Postmenopausal with spontaneous amenorrhea for at least one year, or Spontaneous amenorrhea for more than 6 months and less than one year with Serum Follicular Stimulating Hormone (FSH) level > 40 mIU/mL, or iii. Bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or iv. Total hysterectomy and an absence of bleeding for at least 3 months. 3) BMI: 18.5 to 30.0 kg/m2, both inclusive; BMI value should be rounded off to one significant digit after decimal point (e.g. 30.04 rounds down to 30.0, while 18.95 rounds up to 19.0).

4) Body weight: 50.0 kg to 100.0 kg both inclusive. 5) Able to communicate effectively with study personnel. 6) Willing to provide written informed consent to participate in the study. 7) Judged by the investigator and/or designee to be in good health as documented by the medical history, physical examination (including but may not be limited to an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems), vital sign assessments, 12-lead electrocardiogram (ECG), clinical laboratory assessments, and by general observations. Any abnormalities or deviations outside the normal ranges for any clinical testing (laboratory tests, ECG, etc.) can be repeated at the discretion of the investigator and/or designee and judged to be not clinically significant for study participation. Any abnormalities or deviations outside the normal range for vital signs can be repeated by clinical staff and judged to be not clinically significant for study participation

Exclusion Criteria:

* History of allergic responses to Abatacept or other related drugs, or any of its formulation ingredients.

  2) Any disease or condition which might compromise the haemopoietic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system or any other body system.

  3) History or presence of chronic obstructive pulmonary disease (COPD). 4) Use of any hormone replacement therapy within 3 months prior to the study medication administration.

  5) Use of any depot injection or implant of any drug within 3 months prior to the study medication administration.

  6) Use of CYP enzyme inhibitors or inducers within 30 days prior to the study medication administration (see https://drug-interactions.medicine.iu.edu/MainTable.aspx).

  7) History or evidence of drug dependence. 8) Reports smoking or using tobacco products or is currently using nicotine products (cigarettes, patches, gums, etc.) 14 days prior to screening.

  9) Reports history of drug or alcohol addiction or abuse within the past 1 year.

  10) History of difficulty with donating blood or difficulty in accessibility of veins.

  11) A positive hepatitis screen (hepatitis B surface antigen, hepatitis C antibody).

  12) A positive test result for HIV antibody. 13) A positive QuantiFERON®-TB Gold Plus (Tuberculosis) test. 14) Volunteers who have received a known investigational drug within seven elimination half-lives of the administered drug prior to the study medication administration.

  15) Reports a blood donation totaling between 101 mL to 499 mL within 30 days prior to study drug administration or a blood donation of more than 499 mL within 56 days prior study drug administration for male volunteers and 84 days prior to study drug administration for female volunteers. All volunteers will be advised not to donate blood for 30 days after completing the study.

  16) Intolerance to venipuncture 17) Any food allergy, intolerance, restriction or special diet that, in the opinion of the principal investigator or sub-investigator, could contraindicate the volunteer's participation in this study.

  18) Institutionalized volunteers. 19) Use of any prescribed medications within 14 days prior to the study medication administration.

  20) Use of any OTC products, vitamin and herbal products, etc., within 14 days prior to the study medication administration.

  21) Use of grapefruit and grapefruit containing products within 7 days prior to the study medication administration.

  22) Ingestion of any caffeine or xanthine products (i.e. coffee, tea, chocolate, and caffeine-containing sodas, colas, etc.) for 48 hours prior to administration of study drug, recreational drugs within 30 days prior to screening.

  23) Ingestion of any unusual diet, for whatever reason (e.g.: low sodium) for three weeks prior to the study medication administration.

  24) History of anaphylactic shock. 25) Subjects with current malignancy, history of malignancy, or currently under work-up for suspected malignancy except non-melanoma skin cancer that has been treated or excised and is considered resolved.

  26) Subject has received any live vaccine within one month preceding study drug administration or not able to avoid live vaccines until three months after dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2024-07-04 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter | from baseline till day 70
  Cmax
Pharmacokinetic parameter | from baseline to day 70
  AUCi

SECONDARY OUTCOMES:
Pharmacokinetic parameter | from baseline to day 70
  AUCt
pharmacokinetic parameter | from baseline to day 70
  Tmax
Pharmacokinetic parameter | Baseline to day 70
  T1/2
Pharmacodynamic | basleline to day 70
  ADA (Anti-Drug Antibody) and Neutralizing Anti-drug antibody

CONTACTS AND LOCATIONS:
Overall Officials: Dr Uday Harle, PhD Med, Study Chair — Kashiv Biosciences; Dr Pallav Bharpoda, MBBS, Study Director — Kashiv Biosciences
Locations (1):
- Not Disclosed, Missisauga, Canada